CLINICAL TRIAL: NCT03313141
Title: Study of the Diaphragmatic Function by Transient Elastography : Comparison With Mechanical and Electrophysiological Variables
Brief Title: Study of the Diaphragmatic Function by Transient Elastography (ELASTODIAPH)
Acronym: ELASTODIAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-A00949-40
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: To compare diaphragm elastrography provided by ultrasound to diaphragm function indices provided by magnetic/electrical phrenic nerves stimulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Experimental): Only one arm is considered
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — Volitional and non volitional respiratory tasks
  Other Names: Magnetic and electrical phrenic nerve stimulation

SUMMARY:
The study of diaphragmatic function is usually measured by the pressures and volumes generated by contraction of the diaphragm, which is often difficult (cumbersome technique, difficulty to obtain a perfect cooperation of the subjects, and difficulty to specifically analyze the diaphragm compared to other accessory respiratory muscle groups). In this study, the investigators aimed at analysing diaphragmatic function by measuring the shortening, stiffness, strain and thickening of the diaphragm by ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer

Exclusion Criteria:

* chronic respiratory, neurologic or cardiac disease
* swallowing disorders
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Transdiaphragmatic pressure | 2 hours
  The transdiaphragmatic pressure is the sum of absolute values of gastric and oesophagal pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Pitie Salpêtrière Hospital, Paris, France